CLINICAL TRIAL: NCT04980066
Title: Evaluation of Sticky Bone With or Without EDTA Root Surface Biomodification for Treatment of Gingival Recession: Randomized Controlled Clinical Study
Brief Title: Evaluation of Sticky Bone With or Without EDTA for Treatment of Gingival Recession
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, principal invistigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KD/10/21
Record Dates: First submitted 2021-06-24; First posted 2021-07-28 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Gingival Recession
Keywords: i-PRF; EDTA
MeSH Terms: conditions — Gingival Recession | interventions — Edetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sticky bone and EDTA (Experimental): treatment of gingival recession using sticky bone after root surface biomodification with EDTA
  Interventions: Procedure: Sticky bone and EDTA
- Sticky bone (Active Comparator): treatment of gingival recession using sticky bone
  Interventions: Procedure: Sticky bone

INTERVENTIONS:
Procedure: Sticky bone and EDTA — treatment using Sticky bone after EDTA root surface biomodification
  Arms: sticky bone and EDTA
Procedure: Sticky bone — treatment using Sticky bone
  Arms: Sticky bone

SUMMARY:
Gingival recession is a common clinical finding in periodontal disease which is frequently associated with esthetic concerns, root hypersensitivity, and root caries. Many surgical therapeutic approaches have been developed to predictably obtain root coverage of gingival recession defects. Injectable PRF (I-PRF) is the liquid form of PRF. I-PRF is a bioactive agent obtained by low-speed centrifugation, and it has the capacity to stimulate tissue regeneration. At high concentrations, PRF may stimulate the secretion of several growth factors and trigger fibroblast migration. I-PRF is generally used in regenerative treatments, with good outcomes. Ethylenediaminetetraaceti acid (EDTA) is a chelating agent that could enhance the attachment of connective tissue to the root surface by exposing collagen and, as a consequence, enhance root coverage. EDTA works at neutral pH, and this property has been reported to preserve adjacent tissue vitality. The present study will be carried out to evaluate the effect of sticky bone with or without EDTA root surface biomodification for treatment of gingival recession.

ELIGIBILITY:
Inclusion Criteria:

* Miller I/II isolated maxillary recession defects.
* No abrasion, caries, or cervical restorations and presence of identifiable cementoenamel junction (CEJ).
* No occlusal interferences.
* Full-mouth plaque index (PI) and gingival index (GI) scores of < 1.
* Non-smokers.

Exclusion Criteria:

* Pregnant patients
* Presence of systemic disease or taking medication that interfere with periodontium

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation of root coverage | 6 months
  the percentage of root coverage will be calculated in millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt